CLINICAL TRIAL: NCT07310212
Title: Evaluation of Postoperative Pain and Success Rate Between Lateral Condensation and Warm Vertical Obturation Techniques - A Randomized Controlled Trial
Brief Title: Evaluation of Postoperative Pain and Success Rate Between Lateral Condensation and Warm Vertical Obturation Techniques
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Dalin Al Sawaftah, Endodontic resident, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 224000393
Record Dates: First submitted 2025-08-29; First posted 2025-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Necrotic Pulp; Asymptomatic Apical Periodontitis
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Warm vertical obturation (Active Comparator)
  Interventions: Procedure: Warm Vertical Condensation (WVO)
- Cold lateral condensation obturation (Experimental)
  Interventions: Procedure: Cold Lateral Condensation (CLC)

INTERVENTIONS:
Procedure: Warm Vertical Condensation (WVO) — Following standard endodontic cleaning and shaping with rotary instrumentation and irrigation, canals will be obturated using the warm vertical condensation technique. After placement of a master cone coated with AH Plus sealer, heat is applied to soften and vertically compact the gutta-percha within the canal. The Obtura II system will be used to backfill the canal with thermoplasticized gutta-percha, ensuring three-dimensional adaptation and dense filling of the root canal space.
  Arms: Warm vertical obturation
Procedure: Cold Lateral Condensation (CLC) — Following standard endodontic cleaning and shaping with rotary instrumentation and irrigation, canals will be obturated using the cold lateral condensation technique. A master gutta-percha cone coated with sealer (AH Plus) will be inserted, and accessory cones will be compacted laterally using spreaders until the canal is fully obturated. This technique is widely regarded as the traditional standard method for root canal obturation.
  Arms: Cold lateral condensation obturation

SUMMARY:
Brief Summary

Postoperative pain is a common complication following root canal treatment, particularly in necrotic teeth with asymptomatic apical periodontitis. Although obturation technique has been suggested as a contributing factor to postoperative discomfort, direct clinical comparisons between commonly used methods remain limited. Cold lateral condensation has traditionally been considered the standard obturation technique, while warm vertical obturation systems such as Obtura II have gained popularity due to their potential for improved adaptation of gutta-percha.

This randomized controlled clinical trial aims to compare postoperative pain experience and treatment outcomes following cold lateral condensation and warm vertical obturation in single-rooted necrotic teeth. Postoperative pain will be assessed during the early healing period, along with patient-reported outcomes and short-term clinical and radiographic healing. The results of this study are expected to provide clinically relevant evidence to support evidence-based obturation technique selection and improve patient comfort in endodontic practice.

DETAILED DESCRIPTION:
This study is a prospective, parallel-group randomized controlled clinical trial designed to investigate the influence of obturation technique on postoperative pain experience and short-term treatment outcomes in single-rooted teeth with necrotic pulps.

All endodontic treatments will be performed by a single experienced operator to minimize inter-operator variability. After administration of local anesthesia and placement of rubber dam isolation, standardized access cavities will be prepared. Working length determination will be performed using an electronic apex locator and confirmed radiographically.

Root canal preparation will be carried out using rotary nickel-titanium instruments according to a standardized instrumentation protocol applied uniformly across all participants. Irrigation will be standardized for all cases and will include sodium hypochlorite during instrumentation and ethylenediaminetetraacetic acid (EDTA) for smear layer removal, followed by final canal irrigation and drying using sterile paper points. All procedural steps prior to obturation will be identical between groups to isolate the effect of obturation technique on postoperative outcomes.

Participants will be randomly assigned to one of two obturation techniques:

* Cold lateral condensation, performed using standardized gutta-percha cones and an epoxy resin-based sealer.
* Warm vertical condensation, performed using a thermoplasticized gutta-percha delivery system (Obtura II) in combination with gutta-percha and the same sealer.

Obturation procedures will be conducted according to manufacturer instructions and established clinical guidelines. Immediate coronal sealing will be completed following obturation to reduce the risk of coronal microleakage.

Postoperative pain will be assessed using a Visual Analog Scale (VAS). Participants will receive standardized written and verbal instructions on how to record pain intensity at predefined time points following treatment. Analgesic consumption during the postoperative period will also be documented. Follow-up contact will be made as needed to ensure adherence to pain recording and study protocols.

Clinical and radiographic evaluations will be performed at baseline and at a 6-month follow-up visit to assess treatment outcome and periapical healing. Standardized periapical radiographs will be obtained using consistent exposure parameters. Radiographic assessment will be performed by a blinded assessor to reduce assessment bias.

Randomization will be carried out using sealed opaque envelopes prepared prior to patient recruitment. Due to the nature of the intervention, operator blinding is not feasible; however, patients will be blinded to the obturation technique used, and outcome assessment will be performed by blinded evaluators whenever applicable.

This study is designed to generate controlled clinical evidence regarding the effect of obturation technique on postoperative pain perception and short-term treatment outcomes in necrotic single-rooted teeth, thereby supporting evidence-based clinical decision-making in endodontic practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Patients requiring endodontic treatment for single-rooted necrotic teeth.
* Radiographic and clinical diagnosis of asymptomatic apical periodontitis.
* Ability to understand the study and provide written informed consent.

Exclusion Criteria:

* Teeth diagnosed with symptomatic apical periodontitis.
* Pregnant or lactating women.
* Patients with systemic diseases affecting pain perception (e.g., uncontrolled diabetes, chronic pain conditions).
* Teeth that have been previously endodontically treated.
* Patients taking medications that may influence pain perception (e.g., chronic analgesic or anti-inflammatory drug use).
* Periodontally compromised teeth with significant bone loss or mobility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity following two different obturation techniques | Baseline (6 hours post-treatment), 12 hours post-treatment,1 day, 2 days, 3 days, 4 days, and daily up to 7 days post-treatment
  Visual Analog Scale (VAS), 0-10 0 represents no pain, 10 represents excruciating pain

SECONDARY OUTCOMES:
Patient Satisfaction | Immediately after treatment6 months post treatment
  Questionnaire:
  Extremely satisfied Satisfied Neutral Dissatisfied Extremely dissatisfied
  The maximum is extremely satisfied The minimum is extremely dissatisfied
Assess the need for pain medication | 6 hours post treatment12 hours post treatment1 day2 days3 days4 days up to the complete resolution of pain
  Yes/no
  The check wether or not the patient needed painkillers If yes what time
  'They were advised to take ibupren 400 mg in case of pain and to record when did they need it''
Evaluation of diffrence in success rate | Immediately After treatment 6 months posttreatment
  Comparing Periapical radiographs

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jordan Hospital, Amman, Amman Governate, Jordan

IPD SHARING:
Plan to Share IPD: Undecided